CLINICAL TRIAL: NCT06392100
Title: The Effectiveness of a Mindfulness-Based Intervention in Mental Health, Anxiety, Depression, Stress and Resilience in Generation Z Nursing Students During Clinical Practicum
Brief Title: MBI in Generation Z Nursing Students During Clinical Practicum
Acronym: MBI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Chien Chih-Yin, instructor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MKC-24MMHIS148e
Record Dates: First submitted 2024-04-23; First posted 2024-04-30 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Mental Health; Anxiety; Depression; Resilience
Keywords: Mindfulness-Based Stress Reduction; Generation Z Nursing Students
MeSH Terms: conditions — Psychological Well-Being; Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: The experimental group received mindfulness-based stress reduction intervention, while the control group received weekly line care messages from class instructors. Both groups took the post-test before the internship (T0), during the internship (T1), after the internship (T2), and one month after the internship (T3), a total of 4 times. The contents include psychological well-being scale; anxiety, depression, stress scale and mental toughness scale.
Who Masked: Participant
Masking Description: The experimental group received mindfulness-based stress reduction measures, while the control group received conventional care measures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Intervention in Generation Z Nursing Students During Clinical Practicum (Experimental): The experimental group received mindfulness-based stress reduction intervention for 8 weeks.
  Interventions: Behavioral: Mindfulness-Based Intervention
- line care messages in Generation Z Nursing Students During Clinical Practicum (No Intervention): The control group received line care messages weekly from instructors during clinical practicum.

INTERVENTIONS:
Behavioral: Mindfulness-Based Intervention — Mindfulness-based stress reduction interventions include: breathing awareness, loving-kindness meditation, body scan, walking meditation, sitting body awareness, eating meditation, and deep breathing exercises.
  Other Names: line care messages
  Arms: Mindfulness-Based Intervention in Generation Z Nursing Students During Clinical Practicum

SUMMARY:
This study is a randomized clinical trial design. The research subjects were the internship nursing students in the nursing department of a nursing school in the northern Taiwan.

The experimental group received mindfulness-based stress reduction intervention, while the control group received routine care with weekly line care messages from class instructors. Both groups took the post-test before the internship (T0), during the internship (T1), after the internship (T2), and one month after the internship (T3), a total of 4 times. The contents include psychological well-being scale; anxiety, depression, stress scale and mental scale.

DETAILED DESCRIPTION:
Students need to learn a lot of new medical knowledge and skills during clinical internships, which requires time and effort. However, this kind of learning pressure may put a considerable burden on nursing students, especially anxiety, depression, and stress. Through effective coping strategies, students can improve their confidence in facing clinical situations.

Mindfulness-based stress reduction is a stress-reduction method based on mindfulness meditation. It can relieve the physical and mental stress and anxiety of high-stress people, improve sleep quality, chronic fatigue, and enhance concentration.

The purpose of this study is to explore the effectiveness of mindfulness-based stress reduction intervention on anxiety, depression, and stress in clinical practice of nursing students.

This study adopted a randomized clinical experimental research design. Nursing students from a fifth-level college in the north were selected as the research subjects. A total of 80 people were recruited. Nursing intern students who were willing to participate in the study were randomly assigned and divided into an experimental group of 40 people and a control group. 40 people, the experimental group participated in the mindfulness-based stress reduction course for 8 weeks. The mindfulness-based stress reduction course was led by a certified mindfulness-based stress reduction teacher, once a week, 2 hours each time, for 8 consecutive weeks; the students in the control group received weekly line care messages from the class instructor. Research tools include the General Health Status Scale, Anxiety and Depression Stress Scale, and Mental Resilience Scale. The data were analyzed using SPSS20.0 for Windows.

ELIGIBILITY:
Inclusion Criteria:

* (1) Nursing students during clinical practicum (2) Clear consciousness.

Exclusion Criteria:

-(1) Students diagnosed with schizophrenia, anxiety, depression or affective psychosis.

(2)Taking anti-anxiety medicine treatment or anti-depressant medicine treatment.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Mental Health | Pre-intervention(T0)、Two week after clinical practium begins (T1)、Four week after clinical practium begins(T2)、Two months after clinical practium(T3)
  Psychological Well-Being Scale (PWBS-18) : Ryff & Keyes (1995) proposed that happiness is not only a happy psychological experience, but also a perfect and true performance through one's own efforts. The original scale has 6 facets and 25 questions.
Anxiety, Depression, Stress | Pre-intervention(T0)、Two week after clinical practium begins (T1)、Four week after clinical practium begins(T2)、Two months after clinical practium(T3)
  Depression, Anxiety and Stress Scale - 21 Items (DASS-21)：Developed by scholars at the University of New South Wales in Australia in 1995, it is an internationally authoritative psychological stress assessment tool. It uses a short version of 21 questions to assess common depressive emotions such as depression, anxiety, and stress. There are 21 questions in total, which combine subjective The degree of various induced emotional states is used as an evaluation index, using a 4-point scale, where 1 means not consistent, 2 means sometimes consistent, 3 means usually consistent, and 4 means always consistent.

SECONDARY OUTCOMES:
Resilience | Pre-intervention(T0)、Two week after clinical practium begins (T1)、Four week after clinical practium begins(T2)、Two months after clinical practium(T3)
  Resilience Scale (RS)：The Resilience Scale of Wagnild and Young (1993) focuses on measuring the resilience of individuals at the psychological level, using a seven-point Likert scale with a total of 25 questions.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-yin Chien, master, Study Chair — MacKay Junior College of Medicine, Nursing and Management
Locations (1):
- MacKay Junior College of Medicine, Nursing and Management, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
This study is unwilling to share research data because of confidentiality, privacy protection, legal restrictions, or terms of funding. Additionally, the inability to handle shared data requires additional time and resources to process and manage

REFERENCES:
- [Result] Dong C, Xia L, Zhao C, Zhang X, He J, Zhang G, Zhang J. Prospective association between perceived stress and anxiety among nursing college students: the moderating roles of career adaptability and professional commitment. BMC Psychiatry. 2023 Jun 1;23(1):388. doi: 10.1186/s12888-023-04887-6. PMID 37264378
- [Result] Gurdil Yilmaz S, Yildiz Karadeniz E, dem Lafci D. Clinical-practice stress levels and factors affecting these on first-year nursing students. Perspect Psychiatr Care. 2022 Oct;58(4):3009-3015. doi: 10.1111/ppc.13070. Epub 2022 Mar 22. PMID 35318676
- [Result] O'Driscoll M, Byrne S, Mc Gillicuddy A, Lambert S, Sahm LJ. The effects of mindfulness-based interventions for health and social care undergraduate students - a systematic review of the literature. Psychol Health Med. 2017 Aug;22(7):851-865. doi: 10.1080/13548506.2017.1280178. Epub 2017 Jan 19. PMID 28103700
- [Result] Uysal N, Caliskan BB. The effects of mindfulness-based stress reduction on mindfulness and stress levels of nursing students during first clinical experience. Perspect Psychiatr Care. 2022 Oct;58(4):2639-2645. doi: 10.1111/ppc.13104. Epub 2022 Apr 30. PMID 35488858